CLINICAL TRIAL: NCT01593462
Title: Comparative Effectiveness of MR Enterography, Enteric Ultrasound, and Ultrasound Elastography Imaging in the Evaluation of Pediatric Small Bowel Crohn Disease
Brief Title: Comparative Effectiveness of MR Enterography
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Jonathan R. Dillman M.D., Principal Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00046580
Record Dates: First submitted 2012-04-26; First posted 2012-05-08 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Crohns Disease
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Pediatric Small Bowel Crohn's Disease (Experimental): MRE (magnetic resonance enterography) performed 4 weeks after SBCD treatment begins, or ends or treatment changes, or at 6 months whichever comes first. One research MRE will be performed and one MRE may or may not be performed as part of your routine care.
  Interventions: Procedure: MRE (magnetic resonance enterography); Procedure: The Ultrasound scan, (UEI) Ultrasound Elastography Imaging with ARFI (acoustic radiation force impulse); Behavioral: Study Questionnaires

INTERVENTIONS:
Procedure: MRE (magnetic resonance enterography) — The MRE will take approximately 60 minutes to complete. Enrolled subject will have MRE imaging performed at about 4 weeks after treatment for small bowel crohn's disease begins, and when the treatment ends or changes or at 6 months, whichever comes first. The 4 week MRE will be for research purposes only, the treatment end,change or 6 month MRE may or may not be ordered by the treating physician as part of your routine care. If one is not ordered by the treating physician, the subject will have one performed because of the research study.
Procedure: The Ultrasound scan, (UEI) Ultrasound Elastography Imaging with ARFI (acoustic radiation force impulse) — The US UEI will take about 60 minutes to perform. This exam will be performed by 2 different radiologists and you will have this completed 5 times over the course of the study. This imaging will be performed with the subject drinking oral contrast material. The US, UEI will be completed at baseline, 2 weeks, 4 weeks, 3 months and at treatment end/change or 6 months, whichever comes first.
Behavioral: Study Questionnaires — The subject and their parent will be asked to answer questionnaires 2 weeks after the first MRE and US exams and again after the last imaging examinations are performed at treatment end/change or 6 months, whichever comes first.
  A Pediatric Crohn Disease Activity Index Assessment will be performed at baseline, 2 weeks, 4 weeks, 3 months, and at treatment end/change or 6 months, whichever comes first. The study questionnaires should take no longer than 10 to 40 minutes to complete.

SUMMARY:
The purpose of this study is to determine the efficacy of ultrasound imaging compared to MRE (Magnetic Resonance Enterography) a form of magnetic resonance imaging (MRI) in accurately diagnosing and following Small Bowel Crohn Disease (SBCD) in children.

DETAILED DESCRIPTION:
Computed Tomography (CT) is an imaging tool that exposes patients to radiation, and until recently it was the most commonly used imaging method to evaluate small bowel Crohn disease. Recently, Magnetic Resonance Enterography (MRE) which is a form of magnetic resonance imaging that provides detailed images of the bowel and less frequently, Ultrasound (US) are replacing CT as the standard of care imaging tool at some institutions.

The investigators would like to determine how effective US imaging is compared to MRI imaging in accurately diagnosing and following SBCD in children. Along with enteric ultrasound (EnUS) we will also be comparing a new ultrasound technology called Ultrasound Elastography Imaging (UEI) for this study in which we will be using a second form of UEI called Acoustic Radiation Force Impulse (ARFI). This technique uses sound waves to asses the stiffness properties of soft tissue. The study will compare costs, patient preferences, and imaging accuracy.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric patients under 18 years age.
* Recently diagnosed with small bowel crohn's disease and have not received any prior treatment for this condition

Exclusion Criteria:

* Are pregnant.
* Require sedation to have the MRE exam.
* Cannot tolerate small enclosed spaces for 60 minutes.
* Have kidneys that are poorly functioning (eGFR <30ml/min)

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2011-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Effectiveness of MR Enterography, Enteric US, US Elastography Imaging with ARFI | 6 months
  To assess accuracy in imaging techniques

SECONDARY OUTCOMES:
Cost effectiveness and patient imaging preferences | 6 months
  To compare imaging costs and imaging preferences of the patient.

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Dillman, M.D., Principal Investigator — University of Michigan Hospital; Jonathan Dillman, M.D., Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steien DB, Dillman JR, Lopez MJ, Ehrlich P, Adler J. Morphometric Changes in Children With Small Bowel Crohn Disease During Induction of Therapy: A Pilot Study. J Pediatr Gastroenterol Nutr. 2021 Apr 1;72(4):603-609. doi: 10.1097/MPG.0000000000003009. PMID 33264183